CLINICAL TRIAL: NCT04664023
Title: Description of Immunologic, Enzymatic and Metabolic Biomarkers Associated to the Severity of COVID-19 and Its Resolution
Brief Title: Description of Immunologic, Enzymatic and Metabolic Biomarkers Associated to the Severity of COVID-19 (SARS-CoV-2) and Its Resolution
Acronym: BIOMARK-COVID
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BIOMARK-COVID
Record Dates: First submitted 2020-12-03; First posted 2020-12-11 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Covid19
Keywords: SARS-CoV-2; Immunologic biomarkers; Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood collection at Day 8, Day 16, Day 24, Month 6 and Month 12 after first symptoms from SARS-CoV-2 infection for patients with COVID-19.
  Blood collection at first injection of vaccine against COVID-19, at second injection of vaccine, at Month 1, Month 2, Month 6 and Month 12 after second injection of vaccine for volunteers.
  40mL blood sample will be collected at each blood collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Patients with severe SARS-CoV-2 infection: Patients with severe SARS-CoV-2 infection hospitalised in intensive care unit
  Interventions: Procedure: Blood collection at Day 8, Day 16, Day 24, Month 6 and Month 12 after first symptoms from SARS-CoV-2 infection.
- Patients with intermediate SARS-CoV-2 infection: Patients with intermediate SARS-CoV-2 infection hospitalised in infectious and tropical diseases department
  Interventions: Procedure: Blood collection at Day 8, Day 16, Day 24, Month 6 and Month 12 after first symptoms from SARS-CoV-2 infection.
- Little symptomatic patients with SARS-CoV-2 infection: Little symptomatic ambulatory patients with SARS-CoV-2 infection
  Interventions: Procedure: Blood collection at Day 8, Day 16, Day 24, Month 6 and Month 12 after first symptoms from SARS-CoV-2 infection.
- Patients with SARS-CoV-2 infection hospitalised in geriatry department: Patients with SARS-CoV-2 infection hospitalised in geriatry department to study influence of age on the studied mechanisms
  Interventions: Procedure: Blood collection at Day 8, Day 16, Day 24, Month 6 and Month 12 after first symptoms from SARS-CoV-2 infection.
- Subjects above 65 years wishing to be vaccinated with anti-COVID-19 BioNTech Pfizer vaccine: Subjects above 65 years wishing to be vaccinated with anti-COVID-19 BioNTech Pfizer vaccine
  Interventions: Procedure: Blood collection at 1st injection of vaccine against COVID-19, at at second injection of vaccine, at Month 1, Month 2, Month 6 and Month 12 after second injection of vaccine for volunteers
- Subjects below 65 years wishing to be vaccinated with anti-COVID-19 BioNTech Pfizer vaccine: Subjects below 65 years wishing to be vaccinated with anti-COVID-19 BioNTech Pfizer vaccine
  Interventions: Procedure: Blood collection at 1st injection of vaccine against COVID-19, at at second injection of vaccine, at Month 1, Month 2, Month 6 and Month 12 after second injection of vaccine for volunteers

INTERVENTIONS:
Procedure: Blood collection at Day 8, Day 16, Day 24, Month 6 and Month 12 after first symptoms from SARS-CoV-2 infection. — 40mL blood sample will be collected at each blood collection for immunologic, enzymatic and metabolic biomarker analysis
  Groups: Little symptomatic patients with SARS-CoV-2 infection; Patients with SARS-CoV-2 infection hospitalised in geriatry department; Patients with intermediate SARS-CoV-2 infection; Patients with severe SARS-CoV-2 infection
Procedure: Blood collection at 1st injection of vaccine against COVID-19, at at second injection of vaccine, at Month 1, Month 2, Month 6 and Month 12 after second injection of vaccine for volunteers — 40mL blood sample will be collected at each blood collection for immunologic, enzymatic and metabolic biomarker analysis
  Groups: Subjects above 65 years wishing to be vaccinated with anti-COVID-19 BioNTech Pfizer vaccine; Subjects below 65 years wishing to be vaccinated with anti-COVID-19 BioNTech Pfizer vaccine

SUMMARY:
Prospective study to describe the immunological, metabolic and serologic profile in the acute and post acute phases of Coronavirus disease (COVID-19)

ELIGIBILITY:
Inclusion Criteria for patients:

* adult patient
* Patient with Covid-19 confirmed by RT-PCR, supported by Poitiers hospital
* Patient came for RT-PCR test at the drive of the hospital, or hospitalised in one of the Covid-19 departments of the Poitiers hospital (geriatry, infectious and tropical diseases, medical resuscitation and continuous care unit)
* informed consent signed by the patient or a trusted or immediate person after clear and loyal information on the study

Exclusion Criteria for patients:

* minor patient
* patient having had syptoms for more than 8 days
* patient already enrolled in another study regarding immunomodulators
* patient not benefiting from a Social Security scheme or not benefiting from it through a third party
* patient benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, adult under legal protection

Inclusion Criteria for volunteers:

* adult patient
* subject wishing to be vaccinated with anti-COVID-19 BioNTech Pfizer vaccine
* informed consent signed by the volunteer after clear and loyal information on the study

Exclusion Criteria for volunteers:

* minor patient
* subject having had COVID-19 documented by a positive RT-PCR test or serology
* subject already vaccinated against COVID-19 (complete or partial vaccinal scheme)
* patient not benefiting from a Social Security scheme or not benefiting from it through a third party
* patient benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, adult under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with severe SARS-CoV-2 infection hospitalised in intensive care unit
  Patients with intermediate SARS-CoV-2 infection hospitalised in infectious and tropical diseases department
  Little symptomatic ambulatory patients with SARS-CoV-2 infection
  Patients with SARS-CoV-2 infection hospitalised in geriatry department
  Subjects wishing to be vaccinated with anti-COVID-19 BioNTech Pfizer vaccine
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Neutralizing antibodies | Day 8 following the first SARS-CoV-2 symptoms for patients
  Serum titre of neutralizing antibodies
Neutralizing antibodies | Day 0 of the first injection of vaccine against COVID-19 for volunteers
  Serum titre of neutralizing antibodies
T CD8 lymphocytes | Day 8 following the first SARS-CoV-2 symptoms for patients
  Blood concentration of T CD8 lymphocytes
T CD8 lymphocytes | Day 0 of the first injection of vaccine against COVID-19 for volunteers
  Blood concentration of T CD8 lymphocytes
Inflammatory markers | Day 8 following the first SARS-CoV-2 symptoms for patients
  Blood levels of pro-inflammatory cytokines
Inflammatory markers | Day 0 of the first injection of vaccine against COVID-19 for volunteers
  Blood levels of pro-inflammatory cytokines
Metabolic markers | Day 8 following the first SARS-CoV-2 symptoms for patients
  Blood concentration of glucosidases
Metabolic markers | Day 0 of the first injection of vaccine against COVID-19 for volunteers
  Blood concentration of glucosidases
Neutralizing antibodies | Day 16 following the first SARS-CoV-2 symptoms for patients
  Serum titre of neutralizing antibodies
Neutralizing antibodies | Day 0 of the second injection of vaccine against COVID-19 for volunteers
  Serum titre of neutralizing antibodies
T CD8 lymphocytes | Day 16 following the first SARS-CoV-2 symptoms for patients
  Blood concentration of T CD8 lymphocytes
T CD8 lymphocytes | Day 0 of the second injection of vaccine against COVID-19 for volunteers
  Blood concentration of T CD8 lymphocytes
Inflammatory markers | Day 16 following the first SARS-CoV-2 symptoms for patients
  Blood levels of pro-inflammatory cytokines
Inflammatory markers | Day 0 of the second injection of vaccine against COVID-19 for volunteers
  Blood levels of pro-inflammatory cytokines
Metabolic markers | Day 16 following the first SARS-CoV-2 symptoms for patients
  Blood concentration of glucosidases
Metabolic markers | Day 0 of the second injection of vaccine against COVID-19 for volunteers
  Blood concentration of glucosidases
Neutralizing antibodies | Day 24 following the first SARS-CoV-2 symptoms for patients
  Serum titre of neutralizing antibodies
Neutralizing antibodies | At Month 1 after the second injection of vaccine against COVID-19 for volunteers
  Serum titre of neutralizing antibodies
T CD8 lymphocytes | Day 24 following the first SARS-CoV-2 symptoms for patients
  Blood concentration of T CD8 lymphocytes
T CD8 lymphocytes | At Month 1 after the second injection of vaccine against COVID-19 for volunteers
  Blood concentration of T CD8 lymphocytes
Inflammatory markers | Day 24 following the first SARS-CoV-2 symptoms for patients
  Blood levels of pro-inflammatory cytokines
Inflammatory markers | At Month 1 after the second injection of vaccine against COVID-19 for volunteers
  Blood levels of pro-inflammatory cytokines
Metabolic markers | Day 24 following the first SARS-CoV-2 symptoms for patients
  Blood concentration of glucosidases
Metabolic markers | At Month 1 after the second injection of vaccine against COVID-19 for volunteers
  Blood concentration of glucosidases
Neutralizing antibodies | 6 months following the first SARS-CoV-2 symptoms for patients
  Serum titre of neutralizing antibodies
Neutralizing antibodies | At Month 2 after the second injection of vaccine against COVID-19 for volunteers
  Serum titre of neutralizing antibodies
T CD8 lymphocytes | 6 months following the first SARS-CoV-2 symptoms for patients
  Blood concentration of T CD8 lymphocytes
T CD8 lymphocytes | At Month 2 after the second injection of vaccine against COVID-19 for volunteers
  Blood concentration of T CD8 lymphocytes
Inflammatory markers | 6 months following the first SARS-CoV-2 symptoms for patients
  Blood levels of pro-inflammatory cytokines
Inflammatory markers | At Month 2 after the second injection of vaccine against COVID-19 for volunteers
  Blood levels of pro-inflammatory cytokines
Metabolic markers | 6 months following the first SARS-CoV-2 symptoms for patients
  Blood concentration of glucosidases
Metabolic markers | At Month 2 after the second injection of vaccine against COVID-19 for volunteers
  Blood concentration of glucosidases
Neutralizing antibodies | 12 months following the first SARS-CoV-2 symptoms for patients
  Serum titre of neutralizing antibodies
T CD8 lymphocytes | 12 months following the first SARS-CoV-2 symptoms for patients
  Blood concentration of T CD8 lymphocytes
T CD8 lymphocytes | At Month 6 after the second injection of vaccine against COVID-19 for volunteers
  Blood concentration of T CD8 lymphocytes
Inflammatory markers | 12 months following the first SARS-CoV-2 symptoms for patients
  Blood levels of pro-inflammatory cytokines
Inflammatory markers | At Month 6 after the second injection of vaccine against COVID-19 for volunteers
  Blood levels of pro-inflammatory cytokines
Metabolic markers | 12 months following the first SARS-CoV-2 symptoms for patients
  Blood concentration of glucosidases
Metabolic markers | At Month 6 after the second injection of vaccine against COVID-19 for volunteers
  Blood concentration of glucosidases
Neutralizing antibodies | At Month 12 after the second injection of vaccine against COVID-19 for volunteers
  Blood concentration of glucosidases
T CD8 lymphocytes | At Month 12 after the second injection of vaccine against COVID-19 for volunteers
  Blood concentration of glucosidases
Inflammatory markers | At Month 12 after the second injection of vaccine against COVID-19 for volunteers
  Blood concentration of glucosidases
Metabolic markers | At Month 12 after the second injection of vaccine against COVID-19 for volunteers
  Blood concentration of glucosidases

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.U.de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided